CLINICAL TRIAL: NCT02544022
Title: Development and Validation of Patient Reported Outcome (PRO) Measures for Individuals With Neurofibromatosis 1 (NF1) and Plexiform Neurofibromas (pNFs)
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150195; 15-C-0195
Record Dates: First submitted 2015-09-05; First posted 2015-09-09 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-11-07

CONDITIONS: Neurofibromatosis 1; Plexiform Neurofibromas
Keywords: Pain Scale; QOL; Tool Validation; Cognitive Interviews; Natural History
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1/Phase 1 Focus Group: Patients with NF1 who have PNs and report experiencing pNF related pain and parents of these patients. (completed)
- 2/Phase 1 Patients: Patients with NF1 who have pNFs(completed)
- 3/Phase 1 Parent: Parents of patients in cohort 2 (completed)
- 4/Phase 2 Patients: Patients with NF1 who have pNFs and recent pNF-related pain
- 5/Phase 2 Parents: Parents of patients (ages 8-17 years) enrolled in cohort 4

SUMMARY:
Background:

People with neurofibromatosis 1 (NF1) who have plexiform neurofibromas (pNFs) can have pain that affects their daily lives. This study aims to improve questionnaires that measure their pain, daily living, and physical functioning.

Objectives:

To examine and improve questionnaires about daily living for people with NF1 and pNFs.

Eligibility:

People ages 5 and older with NF1 and a pNF

Design:

Participants will be screened with medical history.

This study will have 2 phases.

Phase 1 participants will talk about existing pain assessment questionnaires and how pNFs affect their life. They will have group discussions of up to 8 people of a similar age with NF1 and pNFs, or the parents of children with it. These will last about 90 minutes. Children ages 5 to 7 and their parents will have one-on-one meetings instead. These will last about 45 minutes. Discussions will be audiotaped. After the questionnaires have been changed, individual interviews will discuss the new wording, instructions, questions, and electronic format of the new forms.

Phase 2 is now complete.

Phase 1 participants may be invited to Phase 2.

Phase 2 participants will complete the new questionnaires. These may be pen-and-paper or electronic. The questionnaires will take about 30 minutes for adults and teens. Children will work one-on-one with a staff member and may need up to 45 minutes. A small group of participants will be complete the forms twice-in clinic and 1 month later at home. Also, a small group who start a new pain treatment or have a dose increase in their treatment will complete the forms twice-before the treatment change and 1 month later.

DETAILED DESCRIPTION:
Background:

* Neurofibromatosis 1 (NF1) is a genetic disease with multiple clinical manifestations, including plexiform neurofibromas (pNFs) that can cause pain and may significantly impact daily functioning and quality of life (QOL).
* Patient-reported outcomes (PROs) are useful in trials for conditions that are disabling and chronic like NF1, where symptom reduction and improved functioning and QOL currently are important treatment outcomes, which may occur with pNF shrinkage.
* A critical step toward approval of drugs to treat pNFs is to evaluate clinical benefit in conjunction with a reduction in tumor volume as assessed by imaging endpoints.
* The FDA requests the use of PROs in NF1 clinical trials, especially for assessing changes in symptoms, such as pain.
* Currently, no valid PRO measures exist that are specific to the NF1 population to assess pNF pain or its functional impact on an individual s life.

Objectives:

* Phase 1: Qualitative Evaluation - COMPLETE

  --To evaluate current modifications and the need for any additional modifications to existing measures of pain intensity (Numeric Rating Scale; NRS-11) and pain interference (Pain Interference Index; PII) and select the most appropriate items to measure physical functioning (PROMIS Physical Functioning; PROMIS-PF) in NF1 based on qualitative feedback from patients with NF1, pNFs and pain to use as endpoints in clinical trials for individuals with NF1 and pNFs.
* Phase 2: Evaluation of Psychometric Properties and Collection of Normative Data
* To evaluate final versions of the NRS-11 (now called the PAin INtensity Scale for pNF [PAINS-pNF]) and PII (now called the Pain Interference Index for pNF [PIIpNF]) measures on reliability, validity, and feasibility in individuals with NF1 and pNFs.

Eligibility:

* Patients with documented NF1 either by NIH clinical criteria or molecularly-proven mutation in the NF1 gene will be included in the study. Patients must have at least 1 plexiform neurofibroma (pNF) that is at least 3cm on longest diameter by physical exam (i.e. visual exam, palpation) or 2D MR imaging OR >=3mL by volumetric MR imaging. Patients must be at least 8 years of age and able to understand, read, and speak English.
* Patients will be ineligible if they were enrolled on a MEK inhibitor trial in the past 12 months or began a new pain treatment regimen (e.g., medication, psychosocial therapy, physical therapy, etc.) within the past three months at the time of recruitment.
* Primary caregivers (i.e. parent, guardian, grandparent) of participants younger than 18 years old are also eligible to participate in order to provide parent report information to further validate the PII-pNF questionnaire for parents.

Design:

* This protocol will be a multi-institutional research study to maximize our ability to assess a large, diverse sample of individuals with NF1.
* This study will consist of 2 phases. During the first phase, we conducted the qualitative portion of the study with individuals with NF1, ages >=5 years, most with pNF-related pain, using both focus groups and individual interviews. During Phase 2, we will evaluate the final electronic versions of the PAINS-pNF and the PII-pNF using a microlongitudinal design to examine internal consistency, construct validity, and test-retest reliability, and to provide normative data on the study measures for the NF1 population.
* Our goal for phase 2 is to recruit between 14 to 16 patients, with a target of 15 in each of the eight phase 2 age bands for an approximate ceiling of 128 patients >=8 years old (target = 120) and 48 parents of children 8-17 years old (target = 45). All patients and parents will be asked to complete the measures two weeks in a row to examine test-retest reliability.

ELIGIBILITY:
* SUBJECT INCLUSION CRITERIA:
* Documented NF1 either by NIH clinical criteria or molecularly-proven mutation in the

NF1 gene, PER the Neurofibromatosis Diagnostic Criteria AND >=1 plexiform neurofibroma in any location that is either symptomatic or asymptomatic, and is defined by the following:

1. a neurofibroma that has grown along the length of a nerve and may involve multiple fascicles and branches OR a spinal neurofibroma that involves two or more levels with connection between the levels or extending laterally along the nerve OR a skin thickness neurofibroma;
2. measures >=3 cm on longest diameter by visual exam, palpation or 2D MR imaging OR >=3 mL by volumetric MR imaging.

   * For phase 1, Age >=5 years. (complete)
   * For phase 2, Age >= 8 years
   * Ability of subject or parent or guardian to understand and the willingness to sign a written informed consent document.
   * Participants must be able to understand, read, and speak the English language.
   * For phase 1 focus groups only, patients need to report experiencing pNF related pain recently with a minimum pain level of 3 on the current NRS-11 or report taking prescription medication that reduces pain and experiencing pNF related pain recently with a minimum pain level of 1 on the current NRS-11. (complete)
   * For phase 2 patients with pain, patients need to report recently experiencing at least a minimal amount of pNF-related pain. Specifically, they will be asked if they recently experienced any pain in a target tumor area and will have to respond yes to be eligible.
   * For phase 2 patients without pain, patients need to report no recent pNF-related pain. Specifically, they will be asked if they recently experienced any pain in a target tumor area and will have to respond no to be eligible.

PRIMARY CAREGIVER INCLUSION CRITERIA:

* Primary caregiver (i.e. parent,guardian, grandparent) who is >= 18 years old of participating subject <= 17 years old
* Participants must be able to understand, read, and speak the English language

EXCLUSION CRITERIA:

* Patients with severe cognitive or behavior impairments who, in the judgment of the investigators, would not be able to cooperate with the study procedures will be excluded.
* Patients cannot be newly enrolled on a clinical trial to treat their pNF or cannot have started a new pain treatment regimen (e.g., medication, psychosocial therapy, physical therapy, etc.) at the time of enrollment. Specifically, patients will be ineligible if they were enrolled on a MEK inhibitor trial in the past 12 months or began a new pain

medication or treatment within the past 3 months prior to enrollment on this study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with documented NF1 either by NIH clinical criteria or molecularly-proven mutation in the NF1 gene will be included in the study. Patients must have at least 1 plexiform neurofibroma (PN) that is at least >3cm on physical exam or >3mL on volumetric MRI. Patients must be at least 5 years of age and able to understand and speak English.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Estimated)
Dates: Start 2015-11-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Realiability | 8 months
  To evaluate final versions of the NRS-11, PII, and PROMIS-PF measures on reliability, validity, sensitivity to change, and feasibility in individuals with NF1 and PNs.
Feasability | 8 months
  To evaluate current modifications and the need for any additional modifications to existing measures of pain intensity (Numeric Rating Scale; NRS-11) and pain interference (Pain Interference Index; PII) and select the most appropriate items to measure physical functioning (PROMIS Physical Functioning; PROMIS-PF) in NF1 based on qualitative feedback from patients with NF1, PNs and pain to use as endpoints in clinical trials for individuals with NF1 and PNs. (completed)

SECONDARY OUTCOMES:
To provide normative data | 8 months
  To provide normative data on these measures of pain intensity and pain interference in individuals with NF1 and pNFs
Convert the measures into electronic format | 8 months
  Convert the measures (including any changes) into an electronic format.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela L Wolters, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (6):
- United States (6):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Cincinnati Children's Hospital and Medical Center Institution, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-C-0195.html